CLINICAL TRIAL: NCT03575091
Title: Physiotherapy Including Frequent Changes of Body Position and Stimulation to Physical Activity for Infants With Bronchiolitis and Other Acute Respiratory Infections - a Randomized Controlled Trial
Brief Title: Physiotherapy for Infants With Bronchiolities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/190
Record Dates: First submitted 2017-10-13; First posted 2018-07-02 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Infant Conditions; Respiratory Insufficiency
Keywords: Infant; Respiration
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Aspiration | interventions — Precision Medicine

STUDY DESIGN:
Intervention Model Description: Comparison of tree parallel groups, 1 control and 2 intervention groups.
Who Masked: Investigator
Masking Description: Randomisation is carried out with sealed envelopes that are only opened just before intervention starts.
  There are different care givers who carry out the observations and who perform the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): The infants will receive the standard care at the ward.
- Non-individualized (Experimental): The parents will be guided manually by the nursing staff and receive written information about how to change body positions of their child regularly throughout the hospital stay.
  Interventions: Other: Non-individualized
- Individualized (Experimental): The infant will receive frequent changes of body positions, stimulation to physical activity, and stimulation to deep breathing while bouncing on a large ball in the arms of an adult. Additional light chest compressions and inhalations may be given. A physiotherapist will perform the intervention at least once daily, and the parents will be manually guided and receive written information about how to change body positions of their child regularly in a similar way throughout the hospital stay.
  Interventions: Other: Individualized

INTERVENTIONS:
Other: Non-individualized — Comparing two experimental interventions with standard care
  Arms: Non-individualized
Other: Individualized — Comparing two experimental interventions with standard care
  Arms: Individualized

SUMMARY:
Children who are in a hospital with respiratory distress often have difficulty breathing, have thick mucus, and may find it hard to eat normally. Sometimes physical therapy is used to treat these children, but it is not entirely known which methods help the children's condition. The aim of this study is to evaluate the most common physiotherapy treatment method that is currently in use in Sweden for infants who are hospitalized with a lower respiratory infection.

DETAILED DESCRIPTION:
All children under 2 years of age who are admitted to the hospital for a respiratory infection and who have previously been essentially healthy are asked to participate. The infants will be randomized to 3 groups, 1 control group and 2 intervention groups. The infants in the control group will receive the standard care at the clinic. In one intervention group the parents will receive instructions how to vary their child body position regularly, and in the other intervention group the child will receive physiotherapy regularly and the parents will carry out some treatment. Further actions in the form of inhalations or stimulation of deep breathing, will be used when needed. The children will be observed following a structured observational protocol regularly throughout the hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Infants hospitalized because of respiratory infections such as bronchiolitis, pneumonia or other airway obstructions.
* Age 0-24 months
* Born in gestation week 35 or later.
* Guardians understand written Swedish, English, Arabic or Persian

Exclusion Criteria:

* Previous cardiac or respiratory disease
* hospitalized more than 24 hours on this occasion

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2018-01-23 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to improvement | Baseline, after 20 minutes, and every third hour up to discharge from hospital, no more than two weeks
  First improvement regarding any of the following: Wang respiratory score, use of supplemented oxygen, use of supplemented high air flow, use of tube feeding, hospital stay

SECONDARY OUTCOMES:
oxygen saturation | Baseline and second assessment, directly following the first intervention (or interval) after 20 minutes
  Change in percutanous oxygen saturation measured by probe on the foot
respiratory rate | Baseline and second assessment, directly following the first intervention (or interval) after 20 minutes
  Change in manually counted RR during one minute
Heart rate | Baseline and second assessment, directly following the first intervention (or interval) after 20 minutes
  Change in pulse oximeter
General condition, parents' assessment | Baseline and every third hour up to discharge from hospital, no more than two weeks
  Time to the first reduction in Numeric Rating Scale 0-10, (0 the best, 10 the worst)
Lung complications | At discharge from the ward, no more than two weeks
  Referral to an intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, PhD, Principal Investigator — Lund University
Locations (2):
- Sweden (2):
  - Skåne University Hospital, Malmo
  - Centrallasarettet, Vaxjo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersson-Marforio S, Lundkvist Josenby A, Hansen C, Ekvall Hansson E. Physiotherapy interventions encouraging frequent changes of the body position and physical activity for infants hospitalised with bronchiolitis: an internal feasibility study of a randomised control trial. Pilot Feasibility Stud. 2022 Mar 30;8(1):76. doi: 10.1186/s40814-022-01030-2. PMID 35351205
- [Derived] Andersson-Marforio S, Lundkvist Josenby A, Ekvall Hansson E, Hansen C. The effect of physiotherapy including frequent changes of body position and stimulation to physical activity for infants hospitalised with acute airway infections. Study protocol for a randomised controlled trial. Trials. 2020 Sep 21;21(1):803. doi: 10.1186/s13063-020-04681-9. PMID 32958026